CLINICAL TRIAL: NCT01707914
Title: Effects of Chinese Bayberry Juice on Liver Enzymes and Plasma Antioxidant Activity in Adult Subjects With Features of Fatty Liver Disease: a Randomised Placebo-controlled Trial
Brief Title: Clinical Investigation on the Effects of Bayberry Juice Treatment in Adult Subjects With Features of Fatty Liver Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shaoguan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: SGU-01; 81172655 (Other Grant/Funding Number: National Natural Science Foundation of China)
Record Dates: First submitted 2012-10-14; First posted 2012-10-16 (Estimated); Last update posted 2012-12-04 (Estimated); Status verified 2012-12

CONDITIONS: Nonalcoholic Fatty Liver Disease
Keywords: oxidative stress; dyslipidemia; inflammation
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Dyslipidemias; Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chinese bayberry juice (Experimental): Consume 500 mL CBJ/d (250 mL CBJ twice daily)
  Interventions: Dietary Supplement: Chinese bayberry juice
- Placebo (Placebo Comparator): Consume 500 mL placebo/d (250 mL placebo twice daily)
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: Chinese bayberry juice — Consume 500 mL CBJ/d (250 mL CBJ twice daily)
  Arms: Chinese bayberry juice
Dietary Supplement: placebo
  Arms: Placebo

SUMMARY:
Chinese bayberry, one of six Myrica species native to China, is rich in anthocyanins, and cyanidin-3-O-glucoside (C3G) was identified as a major anthocyanin component. In previous animal studies from us and other investigators, anthocyanins have been shown to ameliorate dyslipidemia and hepatic steatosis in different rodent models. The aim of the present study was to examine the effects of Chinese bayberry juice (CBJ) on the serum lipid profile and on levels of biomarkers related to antioxidant status in young adults with features of fatty liver disease.

ELIGIBILITY:
Inclusion Criteria:

* Subject inclusion criteria were age 18-25 y,
* BMI [body weight divided by height squared (in kg/m2)] > 23,
* lack of excessive alcohol ingestion confirmed by careful questioning by the primary physician and dietitians (consumption of less than 70 g alcohol in female and 140 g in male per week), and
* the presence of two of the three following diagnostic criteria of the fatty liver disease: increased hepatic echogenicity compared to the spleen or the kidneys, blurring of liver vasculature and deep attenuation of the ultrasonographic signal.

Exclusion Criteria:

* overuse of alcohol,
* viral hepatitis,
* type 1 or 2 diabetes,
* gastrointestinal or connective diseases,
* chronic pancreatitis,
* liver cirrhosis,
* kidney stones, or renal failure;
* use of acetyl-salicylic acid or other antiplatelet drugs, statins of fibrates, oral hypoglycemic drugs, nitrates, nonsteroidal antiinflammatory drugs, corticosteroids, or drugs interfering with coagulation;
* supplementation with vitamins or antioxidants.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2012-06; Primary Completion 2012-10 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Plasma lipids profile | Four weeks

CONTACTS AND LOCATIONS:
Overall Officials: Wenyi Zhong, MD, Study Director — Shaoguan University
Locations (1):
- The affiliated hospital of Shaoguan University, Shaoguan, Guangdong, China

REFERENCES:
- [Derived] Guo H, Zhong R, Liu Y, Jiang X, Tang X, Li Z, Xia M, Ling W. Effects of bayberry juice on inflammatory and apoptotic markers in young adults with features of non-alcoholic fatty liver disease. Nutrition. 2014 Feb;30(2):198-203. doi: 10.1016/j.nut.2013.07.023. PMID 24377455